CLINICAL TRIAL: NCT04539873
Title: Impact of Colchicine in Hospitalized Colombian Patients With COVID-19
Acronym: (COLCOVID19)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: non-inclusion of patients in the study effectively
Sponsor: Fundación Universitaria de Ciencias de la Salud (Other)
Collaborators: Hospital de San Jose (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5175
Record Dates: First submitted 2020-08-29; First posted 2020-09-07 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Corona Virus Infection
Keywords: Colchicine; Gout; Antirheumatic Agents; Tubulin Modulators
MeSH Terms: conditions — Coronavirus Infections; Gout | interventions — Colchicine; Control Groups

STUDY DESIGN:
Intervention Model Description: This is a phase IIIa, prospective, open-label, randomized, parallel-group study designed to evaluate the efficacy and safety of oral colchicine plus standard therapy versus standard therapy in the clinical course of SARS-CoV-2 infection, in a population group with moderate COVID-19 compromise and requiring hospitalization.
  Patients diagnosed with COVID-19 and meeting all eligibility criteria will be randomized for treatment in a 1: 1 ratio through a central voice response system. Randomization will be balanced in each of the 2 strata: 1) hospitalized patients with clinical stage 4 (requirement of supplemental oxygen by nasal contact lenses or mask) of the World Health Organization (WHO) classification, see ANNEX 2, who will receive in addition to the usual treatment for COVID-19 oral colchicine (exposed group); 2) hospitalized patients with clinical stage 4 of the WHO classification who will receive the usual treatment for COVID-19 (control group).
Who Masked: Participant
Masking Description: the sample size of 120 subjects each arm of 60 subjects. Random assignment (1: 1) to either colchicine plus standard treatment or control arm (standard treatment) orally for 14 days. An initial dose of 1.5 mg orally on the first day, followed by 0.5 mg every 12 hours on days 2 to 7 and continuing with 0.5 mg a day until completing 14 days ± 1. It will be followed on days 1, 3, 7, 14, and day 28, evaluating physical examination, clinical situation, laboratories, and adverse events. The primary efficacy data correspond to the deterioration in the clinical status of the patients through the semiquantitative ordinal scale suggested by the WHO R&D committee. Expected results: It is expected to find out how, through different pathways, colchicine could act in modulating or preventing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COLHICINE PLUS STANDARD TREATMENT (Active Comparator): Patients treated in the exposed group will consist of a decreasing dose of colchicine: a dose of 1.5 mg orally on the first day (initial 1 mg and 0.5 mg at 2 hours), followed by 0.5 mg every 12 hours on days 2 to 7, and continuing with 0.5 mg per day until completing 14 ± 1 days. The duration of treatment will be 14 ± 1 days, depending on the clinical judgment of the investigator.
  Interventions: Drug: Colchicine 0.5 MG
- STANDARD TREATMENT (Placebo Comparator): In this case, the centers where the patients will be included adhere to the Colombian guidelines (Colombian Consensus of the Colombian Association of Infectious Diseases), and to standard treatment
  Interventions: Combination Product: CONTROL GROUP

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Patientes in this arm will receive study medication colchicine 1,5 orally on the first day (initially two pills of 0,5 mg and 0.5 mg at 2 hours), followed by 0.5 mg every 12 hours on days 2 to 7, and continuing with 0.5 mg per day until completing 14 ± 1 days. The duration of treatment will be 14 ± 1 days, depending on the clinical judgment of the investigator.
  Other Names: EXPOSED GROUP
  Arms: COLHICINE PLUS STANDARD TREATMENT
Combination Product: CONTROL GROUP — In this case, the centers where the patients are enrolled will adhere to the Colombian guidelines (Colombian Consensus of the Colombian Association of Infectious Diseases)
  Other Names: standard treatment
  Arms: STANDARD TREATMENT

SUMMARY:
This is a phase IIIa, prospective, open-label, randomized, parallel-group study designed to evaluate the efficacy and safety of oral colchicine plus standard therapy versus standard therapy in the clinical course of SARS-CoV-2 infection, in a population group with moderate COVID-19 compromise and requiring hospitalization.Aproximately 120 subjects meeting all inclusion and not inclusion criteria will be randomized to receive either Colchicine plus standard treatment or only standard treatment for 15 days

DETAILED DESCRIPTION:
Introduction: COVID-19 and mortality associated with acute respiratory distress syndrome (ARDS) pose a global public health problem. The increase in spread and associated mortality poses a scenario where cost-effective therapeutic options are urgently and effectively proposed to control and reduce the pandemic and even to reduce the number of deaths Objective: To evaluate the efficacy and safety of oral colchicine plus treatment standard versus standard treatment in the clinical course of SARS-CoV-2 virus infection, in a population group with moderate COVID-19 involvement and requiring hospitalization. Methodology: A prospective, open, randomized, parallel-group study, the sample size of 120 subjects each arm of 60 subjects. Random assignment (1: 1) to either colchicine plus standard treatment or control arm (standard treatment) orally for 14 days. An initial dose of 1.5 mg orally on the first day, followed by 0.5 mg every 12 hours on days 2 to 7 and continuing with 0.5 mg a day until completing 14 days ± 1. It will be followed on days 1, 3, 7, 14, and day 28, evaluating physical examination, clinical situation, laboratories, and adverse events. The primary efficacy data correspond to the deterioration in the clinical status of the patients through the semiquantitative ordinal scale suggested by the WHO R&D committee. Expected results: It is expected to find out how, through different pathways, colchicine could act in modulating or preventing the appearance of ARDS associated with COVID-19, its possible effects on viral replication and antigenic presentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old.
* Laboratory-confirmed SARS-CoV-2 infection: infection confirmed with nasopharyngeal swab by positive RT PCR in the last 48 hours.
* Hospital admission for COVID-19 in the previous 48 hours.
* Clinical stage 3 (no supplemental oxygen requirement) or 4 (supplemental oxygen requirement for nasal contact lenses or mask) of the WHO classification (see ANNEX 2).
* The patient must be able and willing to provide informed written consent before performing study procedures.
* Patient confirmed to covid19 as positive by positive PCR test

Exclusion Criteria:

* Pregnancy, nursing mothers, and women of childbearing potential who are unable to use adequate contraception.
* Known hypersensitivity or other clear contraindication to the use of colchicine.
* History of end-stage renal disease (eGFR <30 ml / min / 1.73 m2).
* Medical history of cirrhosis (Child-Pugh C), liver failure, chronic active hepatitis, or severe liver disease defined by alanine aminotransferase (ALT) or aspartate aminotransferase (AST)> 5 times the upper limit of normal.
* History of pre-existing neuromuscular disease.
* Previous severe hematologic disease or bleeding disorders.
* Inflammatory bowel disease (Crohn's disease or ulcerative colitis), chronic diarrhea, or malabsorptive syndrome.
* Colchicine treatment for other indications.
* Treatment with immunosuppressive/immunomodulatory agents, including glucocorticoids, antivirals, antimalarials, and IL 6 antagonists for 30 days prior to enrollment.
* Use of other investigational drugs at the time of inclusion, or during the 30 days prior to inclusion.
* Any medical condition or disease that, in the opinion of the investigator, may place the patient at unacceptable risk to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who die or require transfer to Intesive care unit | In the first 15 days after ramdomization
  The primary endpoint will be the need of transfert to ICU or composite of dead due to COVID19 infection

SECONDARY OUTCOMES:
Number of participants who die | 15 days after ramdomization
  The secondary end point is the ocurrence of death in the 15 days after ramdomization

CONTACTS AND LOCATIONS:
Overall Officials: JHON JAIME SPROCKEL, MD; IM, Study Chair — Hospital de San Jose
Locations (1):
- Fundación Universitaria de Ciencias de La Salud, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Result] Savarino A, Di Trani L, Donatelli I, Cauda R, Cassone A. New insights into the antiviral effects of chloroquine. Lancet Infect Dis. 2006 Feb;6(2):67-9. doi: 10.1016/S1473-3099(06)70361-9. No abstract available. PMID 16439323
- [Result] Tay MZ, Poh CM, Renia L, MacAry PA, Ng LFP. The trinity of COVID-19: immunity, inflammation and intervention. Nat Rev Immunol. 2020 Jun;20(6):363-374. doi: 10.1038/s41577-020-0311-8. Epub 2020 Apr 28. PMID 32346093